CLINICAL TRIAL: NCT06034821
Title: Rapid Reversal of Suicidal Depression: Comparative Effectiveness of ECT vs. KETAMINE Over the Lifespan (REaKT-SD)
Brief Title: Comparative Effectiveness of ECT vs. KETAMINE Over the Lifespan
Acronym: REaKT-SD
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Johns Hopkins University (Other); University of Pittsburgh (Other); The Cleveland Clinic (Other); Icahn School of Medicine at Mount Sinai (Other); The Center for Addiction and Mental Health (University of Toronto) (Unknown); The University of Texas Health Science Center, Houston (Other); UT Health (Unknown); Mclean Hospital (Other); Massachusetts General Hospital (Other); University of Utah (Other); UC San Francisco (Unknown)
Responsible Party: Principal Investigator, Amit Anand, Professor of Psychiatry, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P001649
Record Dates: First submitted 2023-08-30; First posted 2023-09-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Suicidal Depression (ASD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Subanesthetic dose intravenous ketamine (KET) (Active Comparator): This trial will use standard dose of ketamine (0.5mg/kg infusion over 40 min period) in accordance with research studies that have used ketamine as an antidepressant.
  Interventions: Drug: Subanesthetic dose intravenous ketamine (KET)
- Electroconvulsive therapy (ECT) (Active Comparator): ECT will be given in a standard manner 3 times a week for 4 weeks.
  Interventions: Device: Electroconvulsive therapy (ECT)

INTERVENTIONS:
Drug: Subanesthetic dose intravenous ketamine (KET) — This trial will use standard dose of ketamine (0.5mg/kg infusion over 40 min period) in accordance with research studies that have used ketamine as an antidepressant. Treatments will be given two times a week for a maximum of 8 treatments during the acute arm of the study. The investigators will be able to modify dose and number of treatments as indicated clinically per pragmatic clinical trials procedures. Patients will be clinically assessed prior to each treatment to evaluate response and appropriateness of continuation of treatment. Per FDA guidelines a maximum 60mg/dose will be given regardless of body weight.
  Arms: Subanesthetic dose intravenous ketamine (KET)
Device: Electroconvulsive therapy (ECT) — ECT will be given in a standard manner 3 times a week for 4 weeks. The Initial ECT treatment will be Right Unilateral (RUL) ultra-brief pulse at 6x seizure threshold determined during titration at first visit. If there is not satisfactory improvement with RUL the investigator may change to Bilateral (BL) utilizing brief pulse using 0.5 modified half-age method to determine stimulus intensity. The seizure threshold may increase during the course of treatment and the dose of the electric stimulus may need to be increased incrementally. It is suggested to change to bilateral after three to five RUL treatments if response to treatment is not satisfactory. Treatments will be given three times a week for up to 4 weeks.
  Arms: Electroconvulsive therapy (ECT)

SUMMARY:
This study is a randomized open-label single-blind non-inferiority comparative effectiveness study of ECT vs. KET for the treatment of Acute Suicidal Depression (ASD).

DETAILED DESCRIPTION:
There is a crisis in the treatment of the imminently suicidal patient. Acute Suicidal Depression (ASD) is a life-threatening illness which requires rapid relief. A number of behavioral programs with varying efficacy are available for prevention of suicide. However, once acute suicidal depression has set in, its treatment is woefully inadequate in the current health system despite availability of efficacious treatments. Patients suffering from ASD are usually admitted as inpatients for safety and started on oral antidepressants (which can take 6 - 12 weeks to have an effect) and given nursing care. They are then discharged from the hospital, usually within 4 -5 days, as soon as immediate safety concerns are ameliorated. Essentially, patients do not receive any specific rapidly acting treatment for their suicidal depression. As The immediate post-discharge period has been shown to be of the highest risk for repeat suicide attempts and completed suicides. One important reason for the inadequate treatment of ASD is the lack of large-scale comparative studies of efficacious treatments such as electroconvulsive therapy (ECT) and subanesthetic dose intravenous ketamine (KET). In the absence of data to guide rational treatment choice, neither treatment is being used adequately. Clinicians are less likely to recommend these treatments in the absence of evidence to base their decision regarding which treatment to give first and under what circumstances. Patients are reluctant to choose between these treatments due to uncertainty regarding efficacy and apprehension regarding side effects and social stigma. Finally, in the absence of effectiveness data, hospital administrators and third-party payers are reticent about committing material and financial resources for these services leading to inaccessibility. Hence, there is a critical need for a large-scale comparative effectiveness trial of ECT vs. intravenous ketamine for rapid reversal of ASD to provide rational guidance for all stakeholders.

This study will address this significant clinical dilemma by conducting a large scale (N = 1500) non-inferiority randomized comparative effectiveness trial of ECT vs. KET for rapid treatment of acute suicidal major depression (ASD) across the lifespan.

ELIGIBILITY:
Inclusion Criteria:

1. Considered by a clinician as appropriate for referral to treatment services for rapid reversal of acute suicidal depression.
2. Adults 18 - 90 years of age.
3. Meet DSM-5 criteria for Major Depressive Episode (MDE) as determined by Mini International Neuropsychiatric Interview (MINI PLUS 5.0.0).
4. Acute suicidal ideation or behavior (thinking or behavior suggesting harming or hurting oneself with knowledge that death may result) or attempt (any intentional, non-fatal self-injury regardless of medical lethality, if intent to die was indicated). *
5. Continue to express suicidal ideation since referral as evidenced by Scale for Suicidal Ideation (SSI) ≥6)**
6. Meet the following criteria on symptom rating scales at screening:

   1. Hamilton Depression Scale (HAM-D 17) >15
   2. Montreal Cognitive Assessment (MoCA) of ≥23(to rule out baseline significant cognitive impairment)

Exclusion Criteria:

1. Meeting DSM-5 criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder.
2. Not able to give informed consent to receive ECT or KET treatment.
3. Not able to give informed consent to participate in the study.
4. Meet exclusion criteria for ECT treatment as described in guidelines.
5. Meet exclusion criteria for KET treatment such as:

   1. Pregnant or breast feeding
   2. Satisfying DSM-V criteria of current Mood Depressive Disorder Episode with Psychotic Features (i.e. delusions of hallucinations)
   3. Severe uncontrolled medical illness
   4. Ketamine allergy
6. Intellectual disability and unable to provide consent or follow study procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Scale for Suicidal Ideation (SSI) | Six weeks
  The Scale for Suicidal Ideation (SSI is excellent in terms of test construction and psychometrics (validity and reliability). It has been shown that a SSI score >6 has been found to be predictive of suicide within 6 months of discharge from hospital. At the end of treatment, patients will be assessed for remission of suicidality which is defined as a SSI score <4 i.e. no clinically significant suicidal ideation70. A stringent criterion for remission was chosen as ASD is a life-threatening illness and full remission should be the treatment goal.

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptoms Self Report QIDS-SR | Six weeks
  Self-reported questionnaire
Columbia Suicide Severity Rating Scale (CSSR-S) | 6 weeks
  Clinician rated scales for suicidality and depression
Montgomery Asberg Depression Rating Scale (MADRS) | 6 weeks
  Clinician rated scales
Working Alliance Inventory (WAI-SR) | 6 weeks
  Questionnaire
National Alcohol and Drug Institute (NIDA) Questionnaire | 6 weeks
  Substance use questionnaire
Self and clinician rated scales | 6 weeks
  Measuring length of hospital stay, memory, side effects and quality of life
Brief Psychiatric Rating Scale 4 items (BPRS) | 6 weeks
  4 items for psychosis, higher scores indicate worse outcomes. Range 4-28.
Clinician Administered Dissociative Symptoms Scale (CADSS) | 6 weeks
  Range 0-80, higher scores indicate worse outcomes.
CGI-S | 6 weeks
  Range 1-7, higher scores indicate worse outcomes.
CGI-I | 6 weeks
  Range 1-7, higher scores indicate worse outcomes.
Young Mania Rating Scale (YMRS) | 6 weeks
  Range 0-60, higher scores indicate worse outcomes.
MOCA | 6 weeks
  Range 0-30, higher scores indicate better outcomes.
COWAT (Total words T-score) | 6 weeks
  Range 0-30, higher scores indicate better outcomes.
HVLT-R (Total T-score) | 6 weeks
  Range 0-100, higher scores indicate better outcomes.
IAT | 6 weeks
  Range scores -2-+2
Suicidal Behavior Questionnaire-Revised (SBQ-R) | 6 weeks
  Range 3-18, higher scores indicate worse outcomes.
Global Self Evaluation of Memory (GSE-My) | 6 weeks
  Range 1-7, higher scores indicate worse outcomes.
Patient-rated global assessment of severity and improvement (PGI-S/PGI-I) | 6 weeks
  Range 1-7, higher scores indicate worse outcomes.
Patient Rated Inventory of Side Effects (PRISE) | 6 weeks
  Not scored
Quality of Life Scale (QOLS) | 6 weeks
  Range 16-112, higher scores indicate better outcomes.
Likert Scale Treatment Preference Questionnaire | 6 weeks
  Range 0-7
National Alcohol and Drug Institute (NIDA) substance use questionnaire (TAPS-I and II) | 6 weeks
  Substance specific scores 0-3, higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — Brigham and Woman's Hospital, Harvard Medical School
Locations (10):
- United States (9):
  - UC San Francisco, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UTHealth Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Center for Addiction and Mental Health (University of Toronto), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No